CLINICAL TRIAL: NCT01524250
Title: Recovery of Demyelinating Optic Neuritis After Treatment With Equivalent High Doses of Oral vs. Intravenous Corticosteroids: a Randomized Single Blinded Clinical Trial
Brief Title: Optic Neuritis Recovery After Oral or IV Corticosteroids
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Sarah Morrow, Assistant Professor of Neurology, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB 18804
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Optic Neuritis
Keywords: Multiple Sclerosis; relapse; demyelination; treatment; corticosteroids
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis; Recurrence; Demyelinating Diseases | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral prednisone (Experimental): 1250mg oral prednisone daily for 3 days
  Interventions: Drug: corticosteroids
- IV methylprednisolone (Active Comparator): 1000mg IV methylprednisolone daily for 3 days
  Interventions: Drug: corticosteroids

INTERVENTIONS:
Drug: corticosteroids — 1250mg of oral prednisone daily for 3 days
  Arms: oral prednisone
Drug: corticosteroids — 1000mg IV methylprednisolone daily for 3 days
  Arms: IV methylprednisolone

SUMMARY:
Patients aged 18-65 with acute demyelinating optic neuritis where treatment with high dose corticosteroids are already been chosen by the patient and the diagnosing physician will be contacted for screening and enrollment. Patients will then be randomized to receive equivalent doses of either intravenous (IV) or oral corticosteroid treatment. Optic nerve function assessments will be compared at baseline, prior to treatment, one and six months post corticosteroid treatment. This will allow for a comparison on whether the route of medication plays a role in the effectiveness of treatment with high dose corticosteroids.

DETAILED DESCRIPTION:
This will be a single-blind, randomized comparison study between 1000mg IV methylprednisolone daily for three days and 1250mg oral prednisone daily for three days of the recovery of optic nerve function in acute demyelinating optic neuritis. We will be comparing assessments at baseline, prior to corticosteroid treatment, with assessments at one and six months post corticosteroid treatment.

Patient Population

We propose to study patients with acute demyelinating optic neuritis where treatment with high dose corticosteroids is being considered. This presentation can be either the first presentation of a demyelinating event (CIS) or in a patient with a previous diagnosis of CIS or MS but must be the first presentation of ON in the affected eye.

Subjects will be recruited from out-patients assessed for acute demyelinating optic neuritis by neurology, ophthalmology, neuro-ophthalmology at London Health Sciences Center and St. Joseph's Health Care Center in London, Ontario. Subjects will be included only if the first visit takes place within 14 days of symptom onset. Only subjects where the physician who identifies/diagnoses the optic neuritis is considering corticosteroid treatment will be contacted for potential screening and enrollment. To ensure treatment is chosen based on the clinical judgement of physician diagnosing ON, the investigators will only contact potential subjects after the decision to use corticosteroids has been made by the patient's treating physician.

Primary and Secondary Endpoints

The primary measure will be the P100 latency of the Visual Evoked Potential in the affected eye at six months. Secondary measures will include high contrast visual acuity and contrast sensitivity at one and six months post corticosteroid treatment and the P100 latency at one-month post corticosteroid treatment.

Visual Evoked Potentials VEPs will be recorded with Teca Synergy equipment (Viasys Healthcare). To ensures consistency in technique, the same technician will perform all three assessments (day 0, 30 and 180) on the same patient. The subject's skin will be cleaned for electrode placement. The scalp electrodes will be placed relative to bony landmarks, as per International Society for Clinical Electrophysiology of Vision (ISCEV) standards (40). The electrodes will be positioned 5 cm above the inion for Oz (active), mid-forehead for Fz (reference) and on the right arm for the ground, following ISCEV guidelines. The patient will be positioned comfortably in a chair with the eye at a distance of 1 meter from a 17-inch cathode ray tube (CRT) monitor, which has been found to be superior to an LCD monitor as the latter can cause a delay in the latency. The room will be darkened to minimize extraneous light that produce responses in the visual cortex and interfere with the VEP response. The same room will be used for every VEP in this study. The subject will be monitored for fixation as poor fixation can affect the P100 peak time and an eye patch used to isolate vision from one eye only. Monocular stimulation will occur at a frequency of 2 Hz, beginning with the unaffected eye, averaging 200 individual responses for each trial. A minimum of two trials per eye will be performed as per ISCEV guidelines. Further averaging of additional trials may be done if there are obvious technical problems (with visual fixation for instance). As the test is dependent on subject compliance, the following will take place to maximize compliance and technical aspects of the recording: talking and gum chewing will be prohibited; the subject will be instructed to relax all muscles of the head and neck specifically the jaw; feet will be resting flat on the floor with hands relaxed in the subject's lap; coaching will take place to help diminish any anxiety; the importance of fixation will be emphasized and the need to resist following the changes in colour of the checkerboard pattern and to continue fixating on the red fixation square in the centre of the monitor will be explained. The interpretation of the VEPs will be done by an assessor blinded to the treatment arm received.

Visual Acuity Visual acuity will be measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts and standard protocol as it the gold standard for ophthalmology clinical trials using visual acuity as an outcome. Testing acuity occurs initially at 4 meters initially and only testing at 2 meters if there are no abnormalities noted at 4 meters.

Contrast Sensitivity Contrast sensitivity will be measured using the Low Contrast Sloan Letter Charts that was found to be valid and reliable for the MS population

ELIGIBILITY:
Inclusion Criteria:

1. Males/Females who are ≥ 18 years old and < 65 years old and are capable of understanding and complying with the protocol
2. Have a diagnosis of unilateral acute demyelinating optic neuritis and will be treated with high dose corticosteroids
3. Are within 14 days of symptom onset
4. Have a visual acuity in the affected of eye of ≥ 20/40
5. Have not received corticosteroids in the last thirty (30) days
6. Medications that could potentially affect the VEP P100 amplitude or may cause drowsiness/difficulty with visual fixation are allowed if there has been no change in dose within 30 days of study enrollment or anytime during the study. These medications include:

   1. Carbamazepine or other anticonvulsants (45)
   2. Benzodiazepines
   3. Opioid and opiates
   4. Barbiturates
   5. Sleep aids such as zopiclone or trazadone
   6. Tricyclic antidepressants
7. Have given written informed consent prior to any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his/her future medical care

Exclusion Criteria:

1. Have another medical condition that could affect the visual outcomes, such as, but not limited to, diabetes retinopathy, glaucoma, cataracts and optic neuropathy not due to a demyelinating lesion
2. Have had optic neuritis in the same eye previously

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
P100 latency of the Visual Evoked Potential in the affected eye | 6 months

SECONDARY OUTCOMES:
High contrast visual acuity | one and six months
contrast sensitivity | one and six months
P100 latency of the Visual Evoked Potential in the affected eye | one month

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Center, London, Ontario, Canada

REFERENCES:
- [Derived] Morrow SA, Fraser JA, Day C, Bowman D, Rosehart H, Kremenchutzky M, Nicolle M. Effect of Treating Acute Optic Neuritis With Bioequivalent Oral vs Intravenous Corticosteroids: A Randomized Clinical Trial. JAMA Neurol. 2018 Jun 1;75(6):690-696. doi: 10.1001/jamaneurol.2018.0024. PMID 29507942